CLINICAL TRIAL: NCT06451367
Title: Cardiovascular and Endocrine Response to Muscular Training Program of Young Soccer Players Aged 14-18 Years
Acronym: YoungSoccer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YoungSoccer_14-18
Record Dates: First submitted 2024-05-27; First posted 2024-06-11 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Sport Injury; Hormone Disturbance; Cardiovascular Abnormalities
MeSH Terms: conditions — Endocrine System Diseases; Cardiovascular Abnormalities

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a control group or an intervention group (N=30, with 15 participants in each group). This study focuses on football players aged 14 to 18 who are part of the elite team of the football society of Fribourg, Switzerland.
  In the control group, participants engage exclusively in regular football training, whereas participants in the intervention group also participate in a 12-week neuromuscular development program.
  Measurements
  Before and after the intervention, various measurements are taken for each participant, including:
  Blood steroid profile Heart rate variability Lung function using ergospirometry (VO2 max with lactate) Body composition using the Inbody 770 machine Muscular strength using a Newton measurement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Regular football training and neuromuscular training program for 12 weeks
  Interventions: Other: neuromuscular programm
- Controle (No Intervention): Regular football training

INTERVENTIONS:
Other: neuromuscular programm — neuromuscular programm during 12 weeks (3 times a week, 10 minutes each time)
  Arms: Intervention

SUMMARY:
This study focuses on understanding the cardiovascular and endocrine responses of young soccer players aged 14 to 18 years to a muscular training program. Adolescence is a critical period for physiological development, and investigating these responses can provide insights crucial for athletic performance and overall health. The benefits include promoting overall health, reducing injury risk, and enhancing scientific knowledge. However, intensive training programs may lead to overtraining and potential negative health outcomes if not carefully monitored. The study aims to assess whether additional neuromuscular development over 12 weeks can enhance players' physical fitness and hormonal changes. By examining these outcomes, the study seeks to inform evidence-based training protocols for optimizing adolescent athletes' health and performance in soccer. The study design involves a prospective single-center randomized cohort to investigate these responses comprehensively.

DETAILED DESCRIPTION:
In this study, participants aged 14 to 18, who are part of an elite football team in Fribourg, Switzerland, are randomly assigned to either a control group or an intervention group (N=30, with 15 participants in each group). The control group undergoes regular football training, while the intervention group additionally participates in a 12-week neuromuscular development program. Before and after the intervention, various measurements are taken for each participant, including blood steroid profile, heart rate variability, lung function (VO2 max with lactate), body composition using the Inbody 770 machine, and muscular strength. The control group exclusively engages in regular football training throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Engaging in a football training program.
* No history of injuries in the last 6 months requiring surgical intervention.
* No intake of anabolic supplements.
* Age 14-18 years old.
* Normal BMI (18.5 - 24.9 kg/m²).

Parents and participants must consent to receive all pertinent information discovered during the study, such as potential cardiovascular diseases or hormonal disorders.

Participants must also consent to the sharing of certain private information with their parents or legal guardians. This includes information regarding cannabis use, as well as the consumption of anabolic steroids and other controlled substances. This additional consent ensures transparency and openness in sharing relevant health-related information with parents or legal guardians, particularly for participants under 18 years of age.

For participants under the age of 18, parental consent or consent from a legal guardian is mandatory in addition to the participant's consent. This ensures that minors have parental approval to take part in the study.

All participants, regardless of age, must provide their voluntary consent to participate in the study. For participants under the age of 18, consent from one of their parents or legal guardians is also required in addition to the participant's consent.

Exclusion Criteria:

* Engaging in other supplemental individual exercise programs.
* Being a smoker (>1 cigarette/week).
* Using any medication at the time of testing.
* Having any disease.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-28 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
VO2 max, lactate | Before the start of the 12-week muscular training program (pre-intervention) and immediately after the 12-week intervention (post-intervention).
  The study aims to examine the effects of a 12-week supplemental muscle program on cardiopulmonary exercise testing, focusing on key metrics such as maximum oxygen uptake (VO2max in mL/kg/min with capillary lactate measurement in mmol/L)
Heart rate variability | Before the start of the 12-week muscular training program (pre-intervention) and immediately after the 12-week intervention (post-intervention).
  The study aims to examine the effects of a 12-week supplemental muscle program on cardiopulmonary exercise testing, focusing on key metrics such as heart rate variability (HRV in ms).
Body composition | Before the start of the 12-week muscular training program (pre-intervention) and immediately after the 12-week intervention (post-intervention).
  The study aims to examine the effects of a 12-week supplemental muscle program on cardiopulmonary exercise testing, focusing on key metrics such as body composition (percentage of body fat, muscle mass in kg). Height will be measured in centimeters (cm) and weight in kilograms (kg) to calculate the Body Mass Index (BMI) in kg/m²

SECONDARY OUTCOMES:
Hormonal changes: Cortisol | Before the start of the 12-week muscular training program (pre-intervention) and immediately after the 12-week intervention (post-intervention).
  The study includes a secondary endpoint involving the measurement of cortisol levels (in μg/dL) before and after the muscular training program. These measurements offer valuable insights into the endocrine adaptations induced by the training regimen. By analyzing changes in cortisol levels, researchers can gain a deeper understanding of the hormonal milieu associated with muscle development, recovery, and overall physiological balance.
Hormonal changes: Testosterone | Before the start of the 12-week muscular training program (pre-intervention) and immediately after the 12-week intervention (post-intervention).
  The study includes a secondary endpoint involving the measurement of testosterone levels (in ng/dL) before and after the muscular training program. These measurements offer valuable insights into the endocrine adaptations induced by the training regimen. By analyzing changes in testosterone levels, researchers can gain a deeper understanding of the hormonal milieu associated with muscle development, recovery, and overall physiological balance.

IPD SHARING:
Plan to Share IPD: No